CLINICAL TRIAL: NCT01147510
Title: A Randomized Controlled Study of Montelukast Plus Low Dose Inhaled Budesonide Versus Medium Dose Inhaled Budesonide on Asthma Control in Elderly Patients
Brief Title: Asthma Control in Elderly Patients With Montelukast
Acronym: ACEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Hallym University Medical Center (Other); Wonju Severance Christian Hospital (Other); Korea University Guro Hospital (Other); MCM Vaccines B.V. (Industry)
Responsible Party: Principal Investigator, Hae-Sim Park, Professor, Department of allergy part, Ajou University School of Medicine, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-GEN-CT4-10-095; A070001 (Other Grant/Funding Number: The Korean Health 21 R&D Project and MSD)
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Persistent Asthma; Elderly
Keywords: asthma control in elderly patients; age 60-75
MeSH Terms: interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy of medium dose ICS (Active Comparator)
  Interventions: Drug: Monotherapy of medium dose ICS
- Combination of low ICS and montelukast (Experimental)
  Interventions: Drug: Combination of low ICS and montelukast

INTERVENTIONS:
Drug: Combination of low ICS and montelukast — Two puffs of Pulmicort ® turbuhaler 200µg/puff between 7 a.m. and 10 a.m and take orally a tablet of Singulair® 10mg one time per day.
  Arms: Combination of low ICS and montelukast
Drug: Monotherapy of medium dose ICS — Two puffs of Pulmicort ® turbuhaler 200µg/puff between 7 a.m. and 10 a.m. and between 7 p.m. and 10 p.m. two times per day
  Arms: Monotherapy of medium dose ICS

SUMMARY:
To compare the efficacy of combination therapy of montelukast plus low dose inhaled budesonide and single therapy of medium dose inhaled budesonide on asthma control such as inflammatory markers and clinical indicators and to compare treatment response according to leukotriene related genotypes in elderly patients with asthma

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 - 75 years
* Patients diagnosed with asthma (NIH, 2007) over six months ago
* Patients maintaining monotherapy of low dose inhaled budesonide (pulmicort 400µg/day or ciclesonide 160 µg/day or fluticasone 250 µg/day) or combination of low dose inhaled budesonide and LABA (Seretide® 250 µg/day or Symbicort® 320 µg/day ) for over a month before the participation in this trial
* Patients not reaching 'well controlled asthma status' with four-week monotherapy of low dose inhaled budesonide (Pulmicort 400 µg/day)
* Patients who sufficiently listen to the purpose and content of this trial and the properties of investigational products and voluntarily agree with the participation to sign a written consent approved by IRB of Ajou University Medical Center before the participation in this trial

Exclusion Criteria:

* Patients who show a symptom of an acute disease within 28 days before the beginning of this trial (administration of trial medication)
* Volunteers who are found to be unsuitable through screening tests
* Patients with history of hypersensitivity to montelukast or budesonide
* Patients participating in other clinical trial within three months before the beginning of this trial (administration of trial medication)
* current smokers having more than 10PYs of smoking history
* Patients needing administration of a medication which can affect asthma control such as systemic and immunoregulatory drugs (cyclosporin, omalizumab, etc.) due to a disease except asthma

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Rate of patients reaching "well controlled asthma status" | 12-weeks treatment
  Rate of patients reaching "well controlled asthma status" after 12-week treatment : evaluating comprehensively frequency of day symptoms and night symptoms, limit of activities and use of rescue medicine based on GINA guideline for asthma management (GINA 2006) and PEF or FEV1(% predicted)

SECONDARY OUTCOMES:
Biomarkers of inflammation | baseline(W1), W5, W9, W13, W17
  sputum eosinophils and neutrophils
Time to first well-controlled week | during the 12 weeks of treatment
Sub-group analysis of leukotrienes associated genotypes | visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Sim Park, MD, PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Medical Center, Suwon, South Korea